CLINICAL TRIAL: NCT00251134
Title: OMEGA: A Prospective, Randomised, Double-Blind, Placebo-Controlled Multicentre Study in Patients Who Survived Acute Myocardial Infarction to Investigate the Efficacy and Safety of 1 Gram Ω-3-Fatty Acid Ethyl Esters (Ω-3FAE) Daily Versus Placebo to Reduce the Risk of Sudden Cardiac Death.
Brief Title: OMEGA-Study: Effect of Omega 3-Fatty Acids on the Reduction of Sudden Cardiac Death After Myocardial Infarction
Acronym: OMEGA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Collaborators: Trommsdorff GmbH & Co. KG (Industry); Pronova BioPharma (Industry)
Responsible Party: Prof. Dr. Jochen Senges, Stiftung Institut für Herzinfarktforschung, 67063 Ludwigshafen, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OMEGA
Record Dates: First submitted 2005-11-08; First posted 2005-11-09 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2008-09

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; omega 3-fatty acids
MeSH Terms: conditions — Myocardial Infarction | interventions — zodin; Pharmaceutical Preparations; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): omega-3-acid ethyl ester 90
  Interventions: Drug: Zodin (drug)
- 2 (Placebo Comparator): olive oil
  Interventions: Drug: Olive oil (placebo)

INTERVENTIONS:
Drug: Zodin (drug) — 1 gram omega-3-acid ethyl esters 90 daily for a period of 12 months
  Arms: 1
Drug: Olive oil (placebo) — 1 gram olive oil daily for a period of 12 months
  Arms: 2

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death in North America and Europe. The major cause of CVD is atherosclerosis like coronary artery disease (CAD). The results of recent trials hint that the course of CAD may be positively influenced by an increased intake of omega 3-fatty acids. The OMEGA-Trial analyses this effect in subjects who suffered an acute myocardial infarction. They are divided into two groups, both receiving standard post-infarction therapy. The subjects of one group additionally receive 1 gram of omega 3-fatty acids daily for a time-period of 12 months, while the subjects in the second group receive 1 gram olive-oil as placebo. Within the period of 12 months all events are reported and used to analyse the efficacy and safety of the additional therapy with omega 3-fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial infarction 3-14 days before randomisation (STEMI and NSTEMI)
* Ability to take Ω-3-FAE or olive oil without risk
* Informed consent

Exclusion Criteria:

* Premenopausal women who are not surgically sterile, who are pregnant or nursing, who are of child-bearing potential and are not practising acceptable means of birth control (pregnancy testing required before randomisation)
* Known hypersensitivity to study medication
* Dislike of fish oil
* Haemorrhagic diathesis
* Unwillingness to discontinue other medications containing fish oil
* Legal incapacity
* History of drug or alcohol abuse within 6 months
* Any investigational therapy within one month of signing informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3800 (Actual)
Dates: Start 2003-10; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Sudden cardiac death | 12 months

SECONDARY OUTCOMES:
Total mortality | 12 months
MACCE: Total mortality, re-infarction or stroke | 12 months
Non-fatal resuscitation or survived direct-current (DC)-shock > 30 days | 12 months
Total rehospitalisation | 12 months
Revascularisation: Percutaneous transluminal coronary angioplasty (PTCA) or Coronar artery bypass grafting (CABG) | 12 months
Detection of ventricular tachycardia or fibrillation during 12 months by an ICD, with or without ICD-intervention (shock or antitachycardia pacing). | 12 months
Effect on the severity of depressive co-morbidity in patients surviving an acute myocardial infarction for one year: Mean BDI-II-Depression score and percentage of patients with BDI-II score ≥ 14 | after 12 months
Combined endpoint of Sudden Cardiac Death or adequate ICD-shock/pacing during 12 months | 12 months
Combined endpoint of total mortality or adequate ICD-shock/pacing during 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Senges, Prof. Dr., Principal Investigator — Stiftung Institut fuer Herzinfarktforschung, Chairman
Locations (10):
- Germany (10):
  - Klinikum der Stadt Ludwigshafen gGmbH, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Johanniter-Krankenhaus Rheinhausen, Duisburg
  - Elisabeth-Krankenhaus, Essen
  - Staedt. Kliniken Frankfurt/Main-Hoechst, Frankfurt am Main
  - Klinikum Fuerth, Fürth
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Klinikum Ingolstadt, Ingolstadt
  - Klinikum Neustadt, Neustadt/Aisch
  - Elisabeth-Krankenhaus, Recklinghausen
  - Marienkrankenhaus, Soest

REFERENCES:
- [Background] Rauch B, Schiele R, Schneider S, Gohlke H, Diller F, Gottwik M, Steinbeck G, Heer T, Katus H, Zimmer R, Erdogan A, Pfafferott C, Senges J; Omega-Study Group. Highly purified omega-3 fatty acids for secondary prevention of sudden cardiac death after myocardial infarction-aims and methods of the OMEGA-study. Cardiovasc Drugs Ther. 2006 Oct;20(5):365-75. doi: 10.1007/s10557-006-0495-6. PMID 17124558
- [Derived] Zimmer R, Riemer T, Rauch B, Schneider S, Schiele R, Gohlke H, Diller F, Steinbeck G, Katus H, Senges J; OMEGA-Study Group. Effects of 1-year treatment with highly purified omega-3 fatty acids on depression after myocardial infarction: results from the OMEGA trial. J Clin Psychiatry. 2013 Nov;74(11):e1037-45. doi: 10.4088/JCP.13m08453. PMID 24330904
- [Derived] Rauch B, Riemer T, Schwaab B, Schneider S, Diller F, Gohlke H, Schiele R, Katus H, Gitt A, Senges J; OMEGA study group. Short-term comprehensive cardiac rehabilitation after AMI is associated with reduced 1-year mortality: results from the OMEGA study. Eur J Prev Cardiol. 2014 Sep;21(9):1060-9. doi: 10.1177/2047487313486040. Epub 2013 Apr 4. PMID 23559535
- [Derived] Rauch B, Schiele R, Schneider S, Diller F, Victor N, Gohlke H, Gottwik M, Steinbeck G, Del Castillo U, Sack R, Worth H, Katus H, Spitzer W, Sabin G, Senges J; OMEGA Study Group. OMEGA, a randomized, placebo-controlled trial to test the effect of highly purified omega-3 fatty acids on top of modern guideline-adjusted therapy after myocardial infarction. Circulation. 2010 Nov 23;122(21):2152-9. doi: 10.1161/CIRCULATIONAHA.110.948562. Epub 2010 Nov 8. PMID 21060071